CLINICAL TRIAL: NCT01496794
Title: Prospective Surveillance of Patients With Endophthalmitis for Multi-antibiotic Resistance (PROSPER) Study
Brief Title: Endophthalmitis Cultures
Acronym: PROSPER
Status: Terminated | Type: Observational
Why Stopped: poor enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Stephen J. Kim, MD, Assistant Professor of Ophthalmology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 100487
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Endophthalmitis
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endophthalmitis cultures

SUMMARY:
The intent of this surveillance study will be to obtain written permission from patients with bacterial endophthalmitis in order to compare sterilization rates of their cultured bacterial isolates to standard therapy (vancomycin and ceftazidime) versus combination therapy with vancomycin, ceftazidime, and moxifloxacin.

Research hypothesis:

1. Cultured bacterial isolates will demonstrate faster in vitro sterilization rates with combination treatment (vancomycin, ceftazidime, and moxifloxacin) compared to "standard therapy" with vancomycin and ceftazidime.
2. Longitudinal analysis of resistance patterns of cultured isolates will show increasing rates of multi-antibiotic resistance.

DETAILED DESCRIPTION:
Adult patients over 18 years of age presenting with endophthalmitis and able to sign consent.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients age 18 or greater presenting with bacterial endophthalmitis to the Vanderbilt Eye Institute and who grow positive cultures

Exclusion Criteria:

* Patients < 18 years of age or those patients without positive cultures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vanderbilt Eye Institute
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Kim, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Eye Institute, Nashville, Tennessee, United States